CLINICAL TRIAL: NCT05799248
Title: Role of rhPSMA-7.3 PET/CT Imaging in Men With High-Risk Prostate Cancer Following Conventional Imaging and Associated Changes in Medical Management
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MidLantic Urology (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BED-IIT-437
Record Dates: First submitted 2023-02-21; First posted 2023-04-05 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: role of rhPSMA-7.3 in PET/CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rhPSMA-7.3 (Experimental): Role of rhPSMA-7.3 PET/CT imaging in men with High-Risk prostate cancer following conventional imaging and associated changes in medical management
  Interventions: Drug: rhPSMA-7.3 (18F)

INTERVENTIONS:
Drug: rhPSMA-7.3 (18F) — Patients will receive a dose with an administered activity of 8 mCi (296 MBq) ± 20% of rhPSMA-7.3, delivered as an IV bolus injection with a 10 mL fast 0.9% sodium chloride flush, followed by PET imaging.
  Other Names: radiohybrid PSMA-targeted PET imaging agent, Radioligand for PET CT scanning

SUMMARY:
Study Title: Role of rhPSMA-7.3 PET/CT imaging in men with High-Risk prostate cancer following conventional imaging and associated changes in medical management Protocol number: BED-IIT-437 Phase: 3b Sponsor: MidLantic Urology Funding Organization: Blue Earth Diagnostics Ltd Study Design: This is a Phase 3b, multi-center, single-arm, diagnostic imaging study designed to detect metastatic lesions in men diagnosed with high-risk prostate cancer.

DETAILED DESCRIPTION:
Consented patients will be screened to determine eligibility for the study prior to investigational product (IP) administration. In addition to their routine clinical work-up, which will include 99mtechnetium-biphosphonate bone scan and abdominal/pelvic computed tomography (CT) or magnetic resonance imaging (MRI) and chest CT per local practice, and before the scheduled radical prostatectomy (RP) and pelvic lymph node dissection (PLND), or radical pelvic radiation therapy, patients will receive 8 mCi (296 MBq) ± 20% rhPSMA-7.3, delivered as an intravenous (IV) bolus injection, followed by PET imaging. For each patient, the PET imaging results will be reported to the responsible physician prior to the planned treatment. Imaging results and further procedures/treatment plan should be discussed with the patient within 7 days after rhPSMA-7.3 imaging (this may be conducted by telephone at the clinician's discretion). Within 45 days post-IP administration, the patient will receive treatment as follows:

* Standard of care surgical treatment of PCa, including PLND; or
* If the rhPSMA-7.3 PET scan detects M1 lesion(s):

  * A biopsy/surgery and/or additional imaging to confirm M1 lesion(s) will be required prior to initiation of treatment.

The purpose of this study is to assess the accuracy of rhPSMA-7.3 PET/CT with conventional imaging for detecting metastatic disease in men with high-risk prostate cancer and the impact on medical management of these men. Accurate staging of newly diagnosed PCa assists in directing appropriate treatment strategies. In patients with high-risk PCa, the primary goal of imaging is to detect extra-prostatic disease. The identification of metastatic disease may significantly change the planned treatment regimen from locoregional to systemic therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing to provide signed informed consent and willing to comply with all required study schedule events, where safe and feasible.
2. Patient is male and aged >18 years old.
3. Histologically confirmed adenocarcinoma of the prostate.
4. High risk prostate cancer. High-risk patients will be defined as having any of the following criteria: primary Gleason grade 4, or any Gleason grade 5, PSA ≥20, or clinical stage T3a (per NCCN Guidelines Version 2.2019; PROS-2).

Exclusion Criteria:

1. Patients with any medical condition or circumstance (including receiving an IP) that the investigator believes may compromise the data collected or lead to a failure to fulfil the study requirements.
2. Patients who are planned to have an x-ray contrast agent or other PET radiotracer <24 hours prior to the PET scan.
3. Patients currently receiving, or with a prior history of, androgen deprivation therapy (ADT; defined as surgical orchidectomy; luteinizing hormone-releasing hormone [LHRH] agonist alone [continuous or intermittent]; LHRH antagonist alone [continuous or intermittent]; administration or use of a first generation or second generation anti-androgen alone or in combination with an LHRH agonist/antagonist).
4. Patients participating in an interventional clinical trial within 30 days and having received an IP within five biological half-lives prior to administration of rhPSMA-7.3.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 113 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer upstaging | 15 months
  Compare the accuracy of rhPSMA-7.3 PET/CT with conventional imaging for detecting metastatic disease and up-staging of disease in men with high-risk prostate cancer

SECONDARY OUTCOMES:
Verified Detection Rate of rhPSMA-7.3 | 15 months
  To assess the Verified Detection Rate (VDR) for M1 disease of rhPSMA-7.3 PET/CT findings (as determined by central BIE) on a patient level in with high-risk prostate cancer
Positive predictive value of rhPSMA-7.3 | 15 months
  To assess the VDR and determine PPV for M1 disease of rhPSMA-7.3 PET/CT findings (as determined by central BIE) on a patient level in patients with negative conventional imaging
Metastasis detection rate | 15 months
  Percentage of patients in which rhPSMA-7.3 PET/CT imaging detects at least one verified M1 metastasis, as determined by central BIE
Metastasis detection rate with negative imaging | 15 months
  Percentage of patients with negative conventional imaging for M1 disease in whom rhPSMA-7.3 PET/CT detects at least one verified M1 metastasis, as determined by central BIE
Positive predictive value of rhPSMA compared to biopsy | 15 months
  The PPV of rhPSMA-7.3 PET/CT to detect distant disease compared to biopsy in those patients who undergo a distant disease biopsy on the basis of a rhPSMA-7.3 PET/CT finding or in case of bony disease a correlation with MRI or biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Belkoff, DO, FACOS, Principal Investigator — MidLantic Urology
Locations (1):
- MidLantic Urology, Bala-Cynwyd, Pennsylvania, United States